CLINICAL TRIAL: NCT00513955
Title: A Parallel Randomised Phase II Trial of CHOP Chemotherapy With or Without Bortezomib in Relapsed Mantle Cell Lymphoma
Brief Title: Combination Chemotherapy With or Without Bortezomib in Treating Patients With Relapsed or Refractory Mantle Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital Plymouth NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000559820; NCRN-Ply-26s; EU-20747; ISRCTN200600609024
Record Dates: First submitted 2007-08-08; First posted 2007-08-09 (Estimated); Last update posted 2014-11-05 (Estimated); Status verified 2014-11

CONDITIONS: Lymphoma
Keywords: recurrent mantle cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Mantle-Cell | interventions — Bortezomib; Cyclophosphamide; Doxorubicin; Prednisolone; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bortezomib plus CHOP (Experimental): Patients receive bortezomib IV over 3-5 seconds on days 1 and 8; doxorubicin hydrochloride IV, cyclophosphamide IV, and vincristine IV on day 1; and oral prednisolone on days 1-5.
  Treatment repeats every 21 days for up to 8 courses in the absence of disease progression or unacceptable toxicity.
  Patients complete quality of life questionnaires at baseline, prior to each treatment course, and then at 30 days after completion of treatment.
  After completion of study treatment, patients are followed at 30 days and then every 12 weeks thereafter.
  Interventions: Drug: bortezomib; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: prednisolone; Drug: vincristine sulfate; Other: questionnaire administration; Procedure: quality-of-life assessment

INTERVENTIONS:
Drug: bortezomib
Drug: cyclophosphamide
Drug: doxorubicin hydrochloride
Drug: prednisolone
Drug: vincristine sulfate
Other: questionnaire administration
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as cyclophosphamide, doxorubicin, vincristine, and prednisolone, work in different ways to stop the growth of cancer cells, either by killing the cells or stopping them from dividing. Bortezomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving combination chemotherapy together with bortezomib may kill more cancer cells. It is not yet known whether combination chemotherapy is more effective with or without bortezomib in treating mantle cell lymphoma.

PURPOSE: This randomized phase II trial is studying combination chemotherapy and bortezomib to see how well they work compared with combination chemotherapy alone in treating patients with relapsed or refractory mantle cell lymphoma. Combination chemotherapy alone (Arm I) has been discontinued April 2012 on recommendation of the DMC.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the rates of overall response (complete response [CR], CR unconfirmed [CRu], and partial response).

Secondary

* To evaluate the rates of CR and CRu.
* To determine the median time to progression.
* To determine the median overall survival.
* To evaluate the toxicity and tolerability.
* To compare the responses to these treatment regimens with those from first line therapy.
* To compare the quality of life.

OUTLINE: This is a randomized, open-label, parallel group, multicenter study. Patients are randomized to 1 of 2 treatment arms.

* Arm I (CHOP): Patients receive doxorubicin hydrochloride IV, cyclophosphamide IV, and vincristine IV on day 1 and oral prednisolone on days 1-5. Arm I has been discontinued April 2012 on recommendation of the DMC.
* Arm II (CHOP with bortezomib): Patients receive bortezomib IV over 3-5 seconds on days 1 and 8; doxorubicin hydrochloride IV, cyclophosphamide IV, and vincristine IV on day 1; and oral prednisolone on days 1-5.

In both arms, treatment repeats every 21 days for up to 8 courses in the absence of disease progression or unacceptable toxicity.

Patients complete quality of life questionnaires at baseline, prior to each treatment course, and then at 30 days after completion of treatment.

After completion of study treatment, patients are followed at 30 days and then every 12 weeks thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of mantle cell lymphoma (MCL)

  * Expression of cyclin D1 or evidence of t(11;14) translocation by cytogenetics, FISH, or polymerase chain reaction
* Refractory to or relapsed or progressed after first line antineoplastic therapy
* Measurable disease

PATIENT CHARACTERISTICS:

Inclusion criteria:

* Karnofsky performance status (PS) 50-100% OR ECOG PS 0-2
* ANC ≥ 1,000/mm³ (not related to lymphoma)
* Platelet count ≥ 30,000/mm³
* AST and ALT ≤ 3 times upper limit of normal (ULN)
* Total bilirubin ≤ 2 times ULN
* Creatinine clearance ≥ 20 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

Exclusion criteria:

* Known serological positivity for HBV, HCV, or HIV
* History of allergic reaction attributable to compounds containing boron or mannitol
* Diagnosed or treated for a malignancy other than MCL within the past 5 years except for completely resected basal cell or squamous cell carcinoma of the skin or any in situ malignancy
* Active systemic infection requiring treatment
* Serious medical or psychiatric illness that would preclude study participation

PRIOR CONCURRENT THERAPY:

Inclusion criteria:

* Toxic effects of prior therapy or surgery must be resolved to ≤ grade 2
* Prior splenectomy or localized radiotherapy allowed
* Any prior chemotherapy regimen allowed

  * Chemotherapy may have been given in combination with rituximab
* Concurrent enrollment in a nontreatment study allowed, provided it does not interfere with participation in this study

Exclusion criteria:

* Prior bortezomib
* Antineoplastic therapy within the past 3 weeks
* Nitrosoureas within the past 6 weeks
* Rituximab, alemtuzumab (Campath®), or other unconjugated therapeutic antibody within the past 4 weeks
* Radiotherapy within the past 3 weeks
* Major surgery within the past 2 weeks
* Concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2006-06; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Disease progression | 30 days and every 12 weeks
  The follow-up visits will be at 30 days after last dose of study drug and after that every 12 weeks until: Progressive disease, initiation of further anti-neoplastic therapy, patient decision to withdraw from the study, patient death.
Unacceptable toxicity or tolerability as assessed by NCI CTCAE v3.0 | continual after first drug dose
  The follow-up visits will be at 30 days after last dose of study drug and after that every 12 weeks until: Progressive disease, initiation of further anti-neoplastic therapy, patient decision to withdraw from the study, patient death.

CONTACTS AND LOCATIONS:
Overall Officials: Simon Rule, MD, Study Chair — Derriford Hospital
Locations (25):
- United Kingdom (25):
  - Basingstoke and North Hampshire NHS Foundation Trust, Basingstoke, England
  - Good Hope Hospital, Birmingham, England
  - Birmingham Heartlands Hospital, Birmingham, England
  - Blackpool Victoria Hospital, Blackpool, England
  - Addenbrooke's Hospital, Cambridge, England
  - Darent Valley Hospital, Dartford, England
  - Harrogate District Hospital, Harrogate, England
  - Leeds General Infirmary, Leeds, England
  - Royal Liverpool University Hospital, Liverpool, England
  - Guy's Hospital, London, England
  - Mid Kent Oncology Centre at Maidstone Hospital, Maidstone, England
  - Royal Victoria Infirmary, Newcastle upon Tyne, England
  - James Paget Hospital, Norfolk, England
  - Norfolk and Norwich University Hospital, Norwich, England
  - Derriford Hospital, Plymouth, England
  - Whiston Hospital, Prescot Merseyside, England
  - Southampton General Hospital, Southampton, England
  - Sunderland Royal Hospital, Sunderland, England
  - Musgrove Park Hospital, Taunton, England
  - Torbay Hospital, Torquay, England
  - Royal Cornwall Hospital, Truro, Cornwall, England
  - Aberdeen Royal Infirmary, Aberdeen, Scotland
  - Raigmore Hospital, Inverness, Scotland
  - Ysbyty Gwynedd, Bangor, Wales
  - Prince Philip Hospital, Llanelli, Wales

REFERENCES:
- [Result] Furtado M, Johnson R, Kruger A, Turner D, Rule S. Addition of bortezomib to standard dose chop chemotherapy improves response and survival in relapsed mantle cell lymphoma. Br J Haematol. 2015 Jan;168(1):55-62. doi: 10.1111/bjh.13101. Epub 2014 Aug 22. PMID 25146720